CLINICAL TRIAL: NCT01327456
Title: A Randomized Controlled Trial of a Literacy-sensitive Self-management Intervention for Chronic Obstructive Pulmonary Disease Patients
Brief Title: The Effects of a Self-management Intervention on Low Literacy Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Daniel Jonas, MD / Assistant Professor, University of North Carolina Department of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07-1771
Record Dates: First submitted 2011-03-29; First posted 2011-04-01 (Estimated); Last update posted 2011-04-01 (Estimated); Status verified 2011-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: health literacy; self-management; inhaler technique
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-Management Intervention (Experimental): participants who receive the one-on-one self-management intervention
  Interventions: Behavioral: Self-Management Intervention
- Usual Care (No Intervention): group receives no additional education or intervention then they would as usual care of their COPD

INTERVENTIONS:
Behavioral: Self-Management Intervention — patients will participate in a 1-on-1 interactive intervention, delivered by a trained research assistant targeting self-management skills (e.g. inhaler use, use of an action plan), smoking cessation, and exercise/pulmonary rehabilitation. All participants will return 2-4 weeks after the intervention for a follow-up assessment of inhaler technique use, COPD-related knowledge, and time spent in self-management.
  Arms: Self-Management Intervention

SUMMARY:
Purpose: To determine the role health literacy plays in the care continuum for Chronic Obstructive Pulmonary Disease (COPD) and the effect of a self-management intervention on inhaler technique use, time spent on self-management, and knowledge for COPD patients with low literacy.

Participants: The investigators will recruit patients from the University of North Carolina at Chapel Hill Ambulatory Care Center (ACC) who have a diagnosis of COPD.

Procedures (methods): Potential subjects with COPD will be identified through pharmacy claims data, clinic billing data and the electronic medical record. Eligibility will be prescreened by a research assistant (RA) using the electronic medical record prior to approaching potential subjects for consent. For the first part of the study, consenting subjects will complete a baseline health literacy assessment, a questionnaire, an inhaler technique assessment, and a diary of time spent in self-management activities. Pulmonary function tests (PFT) will be performed on all participants for whom PFTs have not been conducted within the previous 12 months. The questionnaire will include measures of COPD-related knowledge, self-management techniques, quality of care, access, quality of life, costs, healthcare utilization, exacerbations, and basic demographic information. The inhaler technique assessment will be administered by the research assistant using a pre-established protocol. The research assistant will abstract additional data from the medical record to assess the quality of care based on adherence to recommended COPD care guidelines. For the second part of the study, participants will be randomized to control and intervention arms. The self-management intervention will be an interactive experience, delivered by a trained research assistant, targeting self-management skills (inhaler use, using an action plan, etc), smoking cessation, and exercise/pulmonary rehabilitation. Those randomized to the control group will receive usual care. All participants will return 2-4 weeks after the intervention for a follow-up assessment of inhaler technique, COPD-related knowledge, and time spent in self-management.

ELIGIBILITY:
Inclusion Criteria:

* are age 18 years or older and,
* have been diagnosed with COPD
* are active patients in the General Internal Medicine or Pulmonary Clinics at the Ambulatory Care Center
* are being treated with inhaled medication for their COPD

Exclusion Criteria:

* non-English speaking (intervention will be available in English only)
* participants unable to complete the study (either with or without assistance)
* patients who are currently experiencing an exacerbation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
change in Inhaler use technique scores from baseline to follow-up | baseline and at 2-4 weeks later
  The inhaler technique assessment will be conducted by using a pre-established protocol developed to cover the major types of inhalers used by the COPD population. General principles included in the assessment include correct preparation, administration, and if appropriate re-administration of a dose. The assessment will be scored as number of steps completed correctly out of total number of steps assessed.

SECONDARY OUTCOMES:
time spent in self-management activities | 2-4 weeks
  participants will complete a time diary of all COPD related activities
change in COPD-related knowledge from baseline to follow-up | baseline and 2-4 week follow-up
  The baseline questionnaire will include measures of COPD-related knowledge, self-management techniques, quality of care, access to care, quality of life, costs, healthcare utilization, exacerbations, and basic demographic information.
change in smoking status from baseline to follow-up | baseline and 2-4 week follow-up
  assessment of smoking status

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Jonas, MD, Principal Investigator — University of North Carolina; Katie Kiser, Pharm.D., Principal Investigator — University of North Carolina; Darren Dewalt, MD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina Hospitals Ambulatory Care Center, Chapel Hill, North Carolina, United States